CLINICAL TRIAL: NCT01321736
Title: Gut Health Response to a New Fiber Blend
Brief Title: Gut Health Response to Dietary Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1103M96878
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Dietary Fiber
Keywords: dietary fiber; enteral nutrition; laxation
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: dietary fiber — mixture of fiber sources added to liquid nutrition product
  Other Names: mixed fibers include fructans, soluble fiber, and insoluble fiber

SUMMARY:
Dietary fiber is known to influence bowel function. The investigators hypothesize that the addition of a mixture of fibers to liquid diets will improve bowel function as measured by stool weight.

DETAILED DESCRIPTION:
Liquid diets are the sole source of nutrition for many patients. Consumption of liquid diets is linked to lower stool weight. The objective of this study is to feed liquid diets, with and without added fiber, to healthy human subjects to determine if mixed fiber sources can normalize stool weight. Secondary objectives of the study include measurement of gut microbiota and stool chemistry with fiber addition.

ELIGIBILITY:
Inclusion Criteria:

1.Weight

* BMI between 23 - 29
* having obtained his/her informed consent
* willing and able to exclusively consume enteral diets for two 14 day periods
* willing and able to collect stool samples as instructed

Exclusion Criteria:

* any disease
* use of medication except for contraceptive medication and certain OTC medications not affecting laxation
* smoking
* excessive exercise (> 2 hours per week)
* consumption of more than 20 grams of dietary fiber daily
* pregnancy or lactation
* use of laxatives
* use of antibiotics in past 6 months
* use of pre or probiotics supplements in the past 2 months
* use of probiotic foods in the past month
* subjects who cannot be expected to comply with the study procedures
* currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* known allergy or sensitivity to formula ingredients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Stool weight | 5 day collection
  5 day fecal collection on last 5 days of 14 day feeding trial

SECONDARY OUTCOMES:
fecal microbiota | day 14 of feeding trial
  fecal sample on last day of feeding trial will be collected for microbiota analysis

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Koecher KJ, Thomas W, Slavin JL. Healthy subjects experience bowel changes on enteral diets: addition of a fiber blend attenuates stool weight and gut bacteria decreases without changes in gas. JPEN J Parenter Enteral Nutr. 2015 Mar;39(3):337-43. doi: 10.1177/0148607113510523. Epub 2013 Nov 14. PMID 24233256